CLINICAL TRIAL: NCT04458415
Title: The Effect of Traxi Panniculus Retractor on Surgical Time at Non-emergent Cesarean Delivery in Obese Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Collaborator discontinued at this site to pursue the study with a different site.
Sponsor: Geisinger Clinic (Other)
Collaborators: Clinical Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0361
Record Dates: First submitted 2020-06-11; First posted 2020-07-07 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Masking Description: No Masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPR Arm (Experimental): Surgeon will use the Traxi Panniculus Retractor to retract the panniculus during cesarean section.
  Interventions: Other: Traxi Panniculus Retractor (TPR)
- Silk Tape Arm (Active Comparator): Surgeon will use silk tape to retract the panniculus during cesarean section.
  Interventions: Other: Silk Tape

INTERVENTIONS:
Other: Traxi Panniculus Retractor (TPR) — Surgeon uses the Traxi Panniculus Retractor (TPR) surgical retraction device to retract the panniculus during C-Section.
  Arms: TPR Arm
Other: Silk Tape — Surgeon uses silk tape to retract the panniculus during C-Section.
  Arms: Silk Tape Arm

SUMMARY:
This is an unblinded, randomized control trial of obese women to evaluate the impact of the Traxi Panniculus Retractor (TPR) on the cesarean operative time and surgical blood loss when compared to silk tape.

DETAILED DESCRIPTION:
The purpose of the study is to assess whether using the Traxi Panniculus Retractor during cesarean section, in obese (BMI greater than or equal to 30kg/m2 at time of delivery) women, can decrease the cesarean operative time compared to using silk tape to retract the panniculus. Operative time is defined as the time from when the patient lies on the operating room table (at completion of the epidural/spinal anesthesia) until fascial closure.

ELIGIBILITY:
Inclusion Criteria:

* Current BMI equal to or greater than 30 kg/m2 at last prenatal visit or on day of admission to L&D
* Requires panniculus retractor for cesarean delivery, as determined by the surgeon
* Non-emergent cesarean delivery
* Spinal or epidural anesthesia
* Low transverse skin incision
* Gestational age equal to or more than 32 weeks 0 days
* Singleton pregnancy
* Three or less previous cesarean deliveries.
* English speaking

Exclusion Criteria:

* Use of Alexis or any other retractor
* General anesthesia
* Fetal demise
* Placenta previa
* History of bariatric surgery
* Adhesive allergy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Time from when a subject lies on the OR table to fascial closure | During surgery-Time from when a subject lies on the OR table to fascial closure

SECONDARY OUTCOMES:
Time from skin incision to delivery | During surgery-skin incision to delivery
Time from hysterotomy to delivery | During surgery-hysterotomy to delivery
Time from skin incision to closure of fascia | During surgery-skin incision to closure of fascia
Time from skin incision to skin closure | During surgery-skin incision to skin closure

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Paglia, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No